CLINICAL TRIAL: NCT04588675
Title: Assessment of Myocardial Viability by Cardiac Magnetic Resonance Feature Tracking at Rest and During Stress by Low Dose Dobutamine
Brief Title: Stress Cardiac MRI in Ischemic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Emam Eldeen, Principal Investigator, Assiut University
Other Study IDs: Stress cardiac MRI
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — the patients will underwent dobutamine stress cardiac MRI

SUMMARY:
The aim of this study is to assess the diagnostic accuracy of CMR feature-tracking (FT) at rest & during stress with low dose dobutamine (LDD) in the evaluation of viability in ischemic cardiomyopathy (ICM) patients and compare it with delayed gadolinium enhancement (DGE).

ELIGIBILITY:
Inclusion Criteria:

* All patients recruited into the study have chronic LV systolic dysfunction due to coronary artery disease (CAD)

Exclusion Criteria:

* All patients with a contraindication to MR study:

  * Patients with implanted non-MRI compatible electronic devices (e.g. Cardiac pacemakers, intracranial metallic clips, implanted hearing aids, etc.)
  * Patients with foreign bodies in the eye.
  * Claustrophobic patients.
* Patients diagnosed with recent acute coronary syndrome within 4 weeks.
* Patients who had contraindications for MRI or contrast agents, and those with poor image quality due to either inadequate breath holding or arrhythmias

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with chronic LV systolic dysfunction due to coronary artery disease (CAD)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
comparison of myocardial strain with late gadolinium enhancement | Baseline
  analysis of the myocardial strain by low dose dobutamine and test if it can assess myocardial viability

REFERENCES:
- [Background] Bhutani M, Vatsa D, Rahatekar P, Verma D, Nath RK, Pandit N. Role of strain imaging for assessment of myocardial viability in symptomatic myocardial infarction with single vessel disease: An observational study. Echocardiography. 2020 Jan;37(1):55-61. doi: 10.1111/echo.14567. Epub 2019 Dec 23. PMID 31868950
- [Background] Schuster A, Paul M, Bettencourt N, Morton G, Chiribiri A, Ishida M, Hussain S, Jogiya R, Kutty S, Bigalke B, Perera D, Nagel E. Cardiovascular magnetic resonance myocardial feature tracking for quantitative viability assessment in ischemic cardiomyopathy. Int J Cardiol. 2013 Jun 20;166(2):413-20. doi: 10.1016/j.ijcard.2011.10.137. Epub 2011 Nov 29. PMID 22130224